CLINICAL TRIAL: NCT01591668
Title: A Double-Blind, Randomized, Placebo-Controlled, Single and Multiple-Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antiviral Activity of GS-9620 in Treatment Naive Subjects With Chronic Hepatitis C Virus Infection
Brief Title: A Study Evaluating GS-9620 in Treatment Naive Subjects With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-243-0102
Record Dates: First submitted 2012-03-23; First posted 2012-05-04 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis; Hepatitis C; Chronic HCV; HCV; Treatment Naive; Gilead; GS-9620
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 0.3mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose Cohorts GS-9620
- 1mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose Cohorts GS-9620
- 2mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose Cohorts GS-9620
- 4mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose Cohorts GS-9620
- 0.3mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose Cohorts GS-9620
- 1mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose Cohorts GS-9620
- 2mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose Cohorts GS-9620
- 4mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose Cohorts GS-9620

INTERVENTIONS:
Drug: Single Ascending Dose Cohorts GS-9620 — This study will enroll cohorts of 6 eligible, unique subjects per cohort, randomized to either active drug or placebo (5:1) within each cohort. Dose cohorts may be dosed with one of up to 4 possible total weekly doses (0.3 mg, 1 mg, 2 mg, 4 mg). Subjects in Single Ascending Dose (SAD) Cohorts will receive a single dose of GS-9620.
  Arms: 0.3mg GS-9620; 1mg GS-9620; 2mg GS-9620; 4mg GS-9620
Drug: Multiple Ascending Dose Cohorts GS-9620 — This study will enroll cohorts of 6 eligible, unique subjects per cohort, randomized to either active drug or placebo (5:1) within each cohort. Subjects in Multiple Ascending Dose (MAD) Cohorts will receive GS-9620 once weekly for two weeks (QW x 2 doses).
  Arms: 0.3mg GS-9620 QW x 2 doses; 1mg GS-9620 QW x 2 doses; 2mg GS-9620 QW x 2 doses; 4mg GS-9620 QW x 2 doses

SUMMARY:
Dose cohorts may be dosed with one of up to 4 possible total weekly doses (0.3 mg, 1 mg, 2 mg, 4 mg). Dose escalation or repetition will be governed by pre-specified safety and activity rules. Subjects will be confined on either days 1-3 and/or days 8-10. Follow-up visits are also required periodically through day 43. Study procedures involve taking blood samples for pharmacokinetic, pharmacodynamic, virologic, and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18-65 years old
* Chronic HCV infection for at least 6 months, treatment naive
* HCV Viral load > 100,000 IU/mL at Screening
* Monoinfection with HCV 1 genotype
* Hepatitis B surface antigen negative
* Screening ECG without clinically significant abnormalities
* BMI 18-33 kg/m^2
* Creatinine clearing > 70 mL/min
* Negative pregnancy test at screening

Exclusion Criteria:

* Pregnant or lactating subjects
* Co-infection with hepatitis B virus (HBV) or HIV
* History of Gilberts disease
* Particular abnormal laboratory parameters
* Diagnosis of autoimmune disease, poorly controlled diabetes, significant psychiatric illness, severe chronic obstructive pulmonary disease (COPD), malignancy, hemoglobinopathy, retinal disease, and those who are immunosuppressed
* Evidence of hepatocellular carcinoma
* On-going alcohol abuse
* Positive uring drug screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events in single and multiple doses of GS-9620 | Periodically Day 1 to 6 months
  Assessments include adverse events, laboratory abnormalities, 12-lead ECG abnormalities and interval measurements, and vital sign measurements

SECONDARY OUTCOMES:
Assessment of plasma drug concentrations of GS-9620 using non-compartmental methods | Day 1 and Day 8
  Single ascending dose (SAD) cohorts: serial blood samples will be collected on Day 1 at 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, and 96 hours post-dose.
  Multiple ascending dose (MAD) cohorts: serial blood samples will be collected on Day 8 at 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
Measurement of pharmacodynamic markers (cytokines and interferon-stimulated genes [ISGs]) | Days 1, 2, 3, 5, 8
  SAD cohorts: Whole blood and serum for pharmacodynamic (PD) assessments (RNA and cytokine analysis) will be drawn on Day 1: Pre-dose and 8-hour Post-dose, Day 2, Day 3, Day 5, Day 8
  MAD cohorts: Whole blood and serum for PD assessments (RNA and cytokine analysis) will be drawn on Day 1: Pre-dose and 8-hours Post-dose, Day 2, Day 3, Day 5, Day 8: Pre-dose and 8 hours Post-dose, Day 9, Day 10, Day 12, and Day 15
Reduction of hepatitis C (HCV) RNA viral load from baseline | Screening, Baseline, Day 8 or 15
  SAD cohorts: HCV viral load will be drawn at Day 1: Pre-dose, Day 2, 3, 5, 8 and both Follow-up Visits.
  MAD cohorts: HCV viral load will be drawn at Day 1: Pre-dose, Day 2, 3, 5, Day 8: Pre-dose, 9, 10, 15, and both Follow-Up Visits.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Woodland International Research Group, Little Rock, Arkansas
  - Avail Clinical Research, LLC, DeLand, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - CliniLabs, New York, New York
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Alamo Medical Research, San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
- Fundacion De Investigacion De Diego, Santurce, PR, Puerto Rico

REFERENCES:
- [Derived] Lawitz E, Gruener D, Marbury T, Hill J, Webster L, Hassman D, Nguyen AH, Pflanz S, Mogalian E, Gaggar A, Massetto B, Subramanian GM, McHutchison JG, Jacobson IM, Freilich B, Rodriguez-Torres M. Safety, pharmacokinetics and pharmacodynamics of the oral toll-like receptor 7 agonist GS-9620 in treatment-naive patients with chronic hepatitis C. Antivir Ther. 2015;20(7):699-708. doi: 10.3851/IMP2845. Epub 2014 Aug 8. PMID 25105516